CLINICAL TRIAL: NCT04131491
Title: Epilepsy in Alzheimer's Disease: Effect on Disease Progression
Acronym: EADP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UZB-NEU-001
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Mild Cognitive Impairment (MCI) due to AD (Other): Neuropsychological investigation, lumbar puncture, long term-EEG monitoring and/or MEG-EEG, magnetic resonance imaging (MRI), blood sample with deep genetic profiling and Apolipoprotein E (APOE) determination.
  Interventions: Procedure: Lumbar puncture
- Healthy volunteers (Other): Neuropsychological investigation, lumbar puncture, long term-EEG monitoring and/or MEG-EEG, MRI, blood sample with deep genetic profiling and APOE determination.
  Interventions: Procedure: Lumbar puncture

INTERVENTIONS:
Procedure: Lumbar puncture — Lumbar puncture for AD biomarker fluid analysis

SUMMARY:
This is a long-term, prospective, interventional study to investigate the role and prevalence of subclinical epileptiform activity in the hippocampus in patients with mild cognitive impairment (MCI) due to Alzheimer's disease (AD). The investigators would like to investigate whether subclinical epileptiform activity in the hippocampus is more prevalent in patients with MCI, compared to healthy controls and to evaluate its effects on cognitive decline. Evolution of cognitive decline will be assessed over a time period of two years.

DETAILED DESCRIPTION:
Epilepsy is a known comorbidity of Alzheimer's disease. In the past, it was considered to be a late complication of AD. Recent literature suggest seizures to be prevalent much earlier in the time course of the disease. Systematic reviews suggest the occurrence of at least one seizure in 10-22% of AD cases and of epilepsy in 5 out of 100 AD cases. One important factor leading to the underdiagnosis of epilepsy in AD, is the fact that it is difficult to diagnose epilepsy in patients with AD because of an overlap in symptomatology (e.g. speech arrest, staring, confusion, …) A recent pilot study showed that even subclinical epileptiform discharges, without overt epilepsy, were more frequent (42%) in patients with dementia due to AD than in healthy controls (10%). These subclinical epileptic discharges were diagnosed with prolonged electroencephalogram (EEG)-monitoring and magnetoencephalogram (MEG)-registration.

There is overlap in AD and epilepsy pathogenesis. In both diseases, activation of microglia, astrogliosis, neuroinflammation and hippocampal neuronal loss has been described. Studies in mice have shown that hippocampal hyperexcitability is an early electrophysiological impairment in AD, and, that this might be a consequence of soluble Amyloid bèta oligomers. Another study in mice, expressing human Amyloid Precursor Protein (APP), showed hippocampal synchronized large amplitude potentials to be present before onset of spontaneous seizures, memory impairments or Amyloid bèta plaques. Low levels of soluble forms of Amyloid bèta might have increased excitability. Increased neuronal activity per se increases both Amyloid bèta and Tau secretion. This means that recurrent epileptic activity in AD might establish a vicious cycle.

Since hippocampal hyperactivity might be an early electrophysiological impairment in AD according to rodent studies, even before memory impairment exist, the investigators thought it to be useful to track subclinical, hippocampal epileptic activity by use of magnetoencephalogram - high density electroencephalogram (MEG-EEG) in patients with MCI due to AD (aka a stage of predementia) and compare this prevalence to healthy controls. The investigators would also like to track evolution to AD in patients with MCI and subclinical epileptiform activity versus those without.

This could support further investigations, with monitoring of the effect of several antiepileptic drugs in patients with MCI due to AD.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Cognitive concern reflecting a change in cognition reported by patient or informant or clinician
* Objective evidence of impairment in one or more cognitive domains, typically including memory.
* Preservation of independence in functional abilities
* Not demented

Exclusion Criteria:

* Age < 18 years old
* Pregnancy
* Expected death due to illness within 2 years
* Pacemaker or other ferromagnetic material that is not MRI compatible
* Other neurodegenerative or cerebrovascular disease
* Pattern compatible with Normal Pressure Hydrocephalus (NPH) (clinically, imaging)
* Epilepsy
* Multiple sclerosis or other demyelinating disease
* Depression, psychosis or other mental disease
* Use of anti-epileptic drugs
* Alcohol or substance abuse
* Korsakoff syndrome
* Symptomatic liver disease
* Uncontrolled thyroid disorders
* Untreated HIV or syphilis
* Clinically significant vitamin B12 deficiency
* Severe systemic medical illness (eg end-stage cardiac disease, …)

Healthy volunteers Inclusion criteria Age- and gender matched healthy controls

Exclusion criteria

* Age < 18 years old
* Pregnancy
* Pacemaker or other ferromagnetic material that is not MRI compatible
* Mild cognitive impairment or dementia of any cause
* Epilepsy
* Multiple sclerosis or other demyelinating disease
* Depression, psychosis or other mental disease
* Use of anti-epileptic drugs
* Alcohol or substance abuse
* Symptomatic liver disease
* Uncontrolled thyroid disorders
* Untreated HIV or syphilis
* Clinically significant vitamin B12 deficiency
* Severe systemic medical illness (eg end-stage cardiac disease, …)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence, expressed as percentage, of subclinical epileptiform activity in MCI due to AD patients, compared to healthy controls. | Patients will have their investigations at inlcusion within a time frame of 8 weeks. Healthy Volunteers will have their investigations at inclusion within a time frame of 4 weeks.
  Comparison of prevalence of subclinical epileptiform activity (measured by LTM-EEG and MEG)
Odds ratio for conversion to clinical AD when comparing MCI patients with and without subclinical signs of epilepsy at the baseline evaluation. | Patients will have their investigations at inlcusion (time frame: 8 weeks), after 1 year (time frame: 4 weeks) and after 2 years (time frame: 4 weeks).
  Odds ratio of conversion (measured by neuropsychological examination).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nous A, Seynaeve L, Feys O, Wens V, De Tiege X, Van Mierlo P, Baroumand AG, Nieboer K, Allemeersch GJ, Mangelschots S, Michiels V, van der Zee J, Van Broeckhoven C, Ribbens A, Houbrechts R, De Witte S, Wittens MMJ, Bjerke M, Vanlersberghe C, Ceyssens S, Nagels G, Smolders I, Engelborghs S. Subclinical epileptiform activity in the Alzheimer continuum: association with disease, cognition and detection method. Alzheimers Res Ther. 2024 Jan 23;16(1):19. doi: 10.1186/s13195-023-01373-9. PMID 38263073